CLINICAL TRIAL: NCT04042831
Title: A Phase II Study of Olaparib in Patients With Advanced Biliary Tract Cancer With Aberrant DNA Repair Gene Mutations
Brief Title: Olaparib in Treating Patients With Metastatic Biliary Tract Cancer With Aberrant DNA Repair Gene Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-ICRN-1702; NCI-2019-04434 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-ICRN-1702 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2019-07-29; First posted 2019-08-02 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-07

CONDITIONS: Bile Duct Adenocarcinoma; Fanconi Anemia Complementation Group Gene Mutation; Metastatic Bile Duct Carcinoma; PTEN Gene Deletion
MeSH Terms: conditions — Bile Duct Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (olaparib) (Experimental): Patients receive olaparib PO BID on days 1-28. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan or MRI throughout the trial, and collection of blood and tissue samples on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281

SUMMARY:
This phase II trial studies how well olaparib works in treating patients with biliary tract cancer that has spread to other places in the body (metastatic) and with aberrant DNA repair gene mutations. Olaparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy (progression free survival [PFS] rate at first scan) of olaparib monotherapy in advanced biliary tract cancer (BTC) with mutations in deoxyribonucleic acid (DNA) repair genes.

SECONDARY OBJECTIVES:

I. To determine the overall survival of patients with advanced biliary tract cancer with mutations in DNA repair genes treated with olaparib.

II. To determine the progression free survival of patients with advanced biliary tract cancer with mutations in DNA repair genes treated with olaparib.

III. To determine the objective response of patients with advanced biliary tract cancer with mutations in DNA repair genes treated with olaparib.

IV. To assess the duration of response for patients with advanced biliary tract cancer with mutations in DNA repair genes treated with olaparib who experience an objective response.

V. To assess the frequency and severity of adverse events in advanced biliary tract cancer patients treated with olaparib.

CORRELATIVE RESEARCH OBJECTIVES:

I. Determine the prevalence of mutations including those targeting DNA repair pathways.

II. Identify mutational signatures associated with pathogenic process in advanced biliary tract cancer samples.

III. Correlate the presence of mutations and mutational signatures linked to mutations in DNA repair genes and homologous recombinant repair with clinical responses to olaparib.

IV. To evaluate putative biomarkers related to:

Iva. De novo sensitivity. IVb. Tumor evolution and resistance, to PARP inhibition from olaparib in BTC.

OUTLINE:

Patients receive olaparib orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) scan or magnetic resonance imaging (MRI) throughout the trial, and collection of blood and tissue samples on study.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological or cytological documentation of metastatic adenocarcinoma of the biliary tract
* Patients with previously identified genetic aberrations that are associated with homologous recombinant repair pathway will be eligible [e.g. somatic mutations in ATM, ATR, CHEK2, BRCA 1/2, RAD51, BRIP1, PALB2, PTEN, FANC, NBN, EMSY, MRE11, ARID1A] or germline mutations in the above genes. Clinical Laboratory Improvement Act (CLIA)-certified assays including commercial tests (Foundation Medicine, Caris, Tempus) will be allowed
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2. (Form is available on the Academic and Community Cancer Research United [ACCRU] website)
* Life expectancy of >= 16 weeks per estimation of investigator
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 7 days prior to registration)
* Platelet count >= 75,000/mm^3 (obtained =< 7 days prior to registration)
* Hemoglobin >= 9.0 g/dL with no blood transfusion in the past 28 days (obtained =< 7 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 7 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer) (obtained =< 7 days prior to registration)
* Serum creatinine =< 1.5 x ULN (obtained =< 7 days prior to registration)
* Institutional normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN (obtained =< 7 days prior to registration)

  * Exception: Patients who are therapeutically treated with anticoagulant agents will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care
* Alkaline phosphatase limit =< 2.5 x ULN (=< 5 x ULN for patients with liver involvement of their cancer) (obtained =< 7 days prior to registration)
* Creatinine clearance estimated of >= 51 mL/min using the Cockcroft-Gault equation (obtained =< 7 days prior to registration)
* Negative serum pregnancy test done =< 28 days prior to registration and confirmed prior to treatment on day 1, for women of childbearing potential, postmenopausal women or women of childbearing potential with evidence of non-childbearing status.

  * Postmenopausal is defined as:

    * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
    * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50
    * Radiation-induced oophorectomy with last menses > 1 year ago
    * Chemotherapy-induced menopause with > 1 year interval since last menses
    * Surgical sterilization (bilateral oophorectomy or hysterectomy)
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide blood and tissue for correlative purposes
* Hepatitis B virus surface antigen (HBsAg), anti-hepatitis B virus core antigen (anti-HBc) and hepatitis B virus surface antigen (anti-HBs)
* Patients with chronic HBV receiving any systemic anticancer therapy should receive antiviral prophylactic therapy through and for minimum 12 months following anticancer therapy
* Patients with past HBV undergoing other systemic anticancer therapies not clearly associated with a high risk of HBV reactivation should be monitored with HBsAg and alanine aminotransferase during cancer treatment (suggest every other cycle)

Exclusion Criteria:

* Platinum refractory disease which was defined as:

  * Evidence disease progression on platinum based chemotherapy regimen or
  * Evidence of disease progression =< 6 months of completion of platinum based adjuvant chemotherapy regimen
* Patient has received prior systemic anti-cancer therapy, tumor embolization or radiotherapy =< 28 days prior to registration
* Major surgical procedure, open biopsy, or significant traumatic injury =< 28 days prior to registration

  * NOTE: Patients must have recovered from any effects of any major surgery
* Congestive heart failure - New York Heart Association (NYHA) >= class II
* Resting electrocardiogram (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg. unstable ischemia, uncontrolled symptomatic arrhythmia, corrected QT interval by Fridericia's correction formula [QTcF] prolongation > 500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome. Cardiac arrhythmias requiring anti-arrhythmic therapy.

  * NOTE: Pacemaker, beta blockers or digoxin are permitted
* Uncontrolled hypertension - grade 3 or higher per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. (despite optimal medical management)
* History of or current pheochromocytoma
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism =< 6 months prior to registration
* Ongoing infection > grade 2 National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0
* Seizure disorder requiring medication
* Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has a negative imaging study =< 28 days of registration and is clinically stable with respect to the tumor at the time of registration. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days prior to registration

  * NOTE: The patient can receive a stable dose of corticosteroids before and during the study as long as these were started =< 28 days prior to registration
* History of organ allograft (including corneal transplant) or allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Evidence or history of bleeding diathesis or any hemorrhage or bleeding event > CTCAE v5.0 grade 3, =< 28 days prior to registration
* Non-healing wound, ulcer, or bone fracture
* Renal failure requiring hemo-or peritoneal dialysis
* Dehydration CTCAE v5.0 grade >= 2
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* Persistent proteinuria of CTCAE v5.0 grade 3 or higher (>= 3.5 g/24 hours [hrs])
* Unable to swallow orally administered medications
* Any malabsorption condition and/or patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Unresolved toxicity greater than CTCAE v5.0 grade 2 attributed to any prior therapy/procedure excluding alopecia and oxaliplatin induced neurotoxicity =< grade 2
* Albumin levels < 2.5 g/dl
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown.

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
  * NOTE: Women of childbearing potential and their partners, who are sexually active, must agree to the use of TWO highly effective forms of contraception in combination. This should be started from the time of registration and continue throughout the period of taking study treatment and for at least 1 month after last dose of study drug(s), or they must totally/truly abstain from any form of sexual intercourse.
  * Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential. Male patients should not donate sperm throughout the period of taking olaparib and for 3 months following the last dose of olaparib
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) serologically positive and currently receiving antiretroviral therapy.

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Previous and/or intercurrent cancers. With the exception of: curatively-treated cancers with no recurrence in >= 5 years or early cancers treated with curative intent, including but not limited to cervical carcinoma in situ, superficial, noninvasive bladder cancer, basal cell carcinoma, squamous cell carcinoma in situ, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, or endoscopically resected gastrointestinal cancers limited in mucosal layer

  * NOTE: All cancer treatments for cancers that were distinct in a primary site other than biliary tract cancer must be completed >= 3 years prior to registration
* Pleural effusion or ascites that causes respiratory compromise (>= CTCAE v5.0 grade 2 dyspnea)
* Previous enrollment in the present study
* Prior exposure to any PARP inhibitor including olaparib
* Known hypersensitivity reaction to olaparib or any of the excipients of the product
* Myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of myelodysplastic syndrome/acute myeloid leukemia (MDS/AML)
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil).

  * NOTE: The required washout period prior to registration is 2 weeks
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil).

  * NOTE: The required washout period prior to registration is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
* Patient taking medications or herbal products including grapefruits, grapefruit hybrids, pomelos, star fruits, Seville oranges, pomegranates, or the juice from any of these. Note: Patients must discontinue the drug/product >= 7 days prior to registration
* Patient taking medications with a known risk to prolong the QTc interval and/or cause Torsades de Pointes. Note: Patients must be discontinued >= 7 days of registration. Treating physicians may wish to replace the drug(s) that do not carry this risk with safe alternative(s)
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable outside of 28 days prior to treatment)
* Involvement in the planning and/or conduct of the study
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) at first scan | At first scan (approximately 8 weeks)
  A patient is defined as a success if the patient is progression-free and alive at the first disease evaluation scan. Disease status will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria. The PFS rate will be calculated as the proportion of evaluable patients who are progression-free and alive at the first disease assessment scan. The final PFS rate point estimate and corresponding 95% confidence interval (CIs) will be reported according to the method of Clopper-Pearson.

SECONDARY OUTCOMES:
Overall survival (OS) | From study entry to death from any cause, assessed up to 3 years
  Patients who are still alive at the time of analysis will be censored at the time of their last study assessment (if still actively on the study) or at the date, the patient was last known to be alive (if in survival follow-up). OS will be estimated using the Kaplan-Meier method. The median OS and corresponding 95% confidence interval (by Brookmeyer and Crowley) will be reported.
PFS | From study entry to the first of either disease progression or death from any cause, assessed up to 3 years
  Progression free survival is defined as the time from study registration to disease progression or death, whichever occurs first. Disease progression will be determined based on RECIST 1.1 criteria. Patients who do not experience disease progression or death while on the protocol will be censored at their last disease assessment date. PFS will be estimated using the Kaplan-Meier method. Median PFS and corresponding 95% CIs (by Brookmeyer and Crowley) will be reported.
Objective response rate | Up to 3 years
  Objective response (unconfirmed) is defined as achieving a complete or partial response while on treatment. The objective response rate (ORR) will be calculated as the proportion of evaluable patients who achieve an objective response. Disease status will be assessed using RECIST v1.1 criteria. Confidence intervals for the true success proportion will be calculated according to the approach of Clopper and Pearson.
Duration of response (DoR) | Up to 3 years
  Will be defined for all evaluable patients who have achieved an objective response as the date at which the patient's earliest best objective status is first noted to be either a complete response or partial response to the earliest date progression is documented, or death if no prior evidence of disease progression. The distribution of DoR will be estimated using the method of Kaplan-Meier. The median DoR and corresponding 95% confidence interval will be reported.
Incidence of adverse events | Up to 3 years
  Adverse events by patients will be summarized by frequencies and severity using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The proportion of patients who experience at least one grade 3+ adverse event (regardless of attribution) will be reported.

OTHER OUTCOMES:
Prevalence of mutations | Up to 3 years
  Will determine the prevalence of mutations including those targeting DNA repair pathways.
Mutational signatures | Up to 3 years
  Will identify mutational signatures associated with pathogenic process in advanced biliary tract cancer samples. Genomic analyses will be performed on mandatory blood samples collected from patients at the start of therapy, every 8 weeks, and at progression.
Presence of mutations and mutational signatures | Up to 3 years
  Will correlate the presence of mutations and mutational signatures linked to mutations in DNA repair/HRR with clinical responses.
The number of patients that had biomarkers related to de novo sensitivity | Up to 3 years
  Will evaluate putative biomarkers related to: (a) de novo sensitivity and (b) tumor evolution and resistance, to PARP inhibition in biliary tract cancer.
  related to: (a) de novo sensitivity and (b) tumor evolution and resistance, to PARP inhibition in BTC.
The number of patients that had biomarkers related to tumor evaluation and resistance | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Ahn, Principal Investigator — Academic and Community Cancer Research United
Locations (6):
- United States (6):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas